CLINICAL TRIAL: NCT01092650
Title: Determining Levels of [D10] Phenanthrene Tetraol in Smokers' Urine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0707M13481
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Tobacco Toxicant Exposure
Keywords: Tobacco toxicants; Polycyclic aromatic hydrocarbons; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Smoked (Active Comparator): Deuterated Phenanthrene spiked in a study cigarette
  Interventions: Drug: Deuterated phenanthrene
- Oral (Experimental): Deuterated phenanthrene in an oral dose
  Interventions: Drug: Deuterated phenanthrene

INTERVENTIONS:
Drug: Deuterated phenanthrene — Deuterated phenanthrene 10 micrograms

SUMMARY:
The purpose of this research study is to better understand how people respond to cancer-causing chemicals in cigarette smoke. Some people are able to get rid of these chemicals as harmless agents while others suffer damage to their cells that can ultimately result in cancer. We hope to develop a better understanding of how we can identify the people who are in danger of getting cancer. Participants will complete questionnaires regarding their health and smoking history. We will take blood samples to look at genes which determine how the body breaks down some tobacco-related toxins. Participants will be given a small amount of liquid to drink, containing alcohol, water, and a compound called deuterated phenanthrene (DP), which is found in cigarette smoke and in the environment. Phenanthrene is non-toxic and does not cause cancer, but this compound is broken down by the body in the same way as cancer-causing agents. We will follow the pathway of this compound as it is broken down in the body.

DETAILED DESCRIPTION:
Forty apparently healthy smokers and non smokers (20 male, 20 female) will be recruited by advertising in the Twin Cities area. This will be done by the Tobacco Use Research Center. They will be screened in a phone call, then invited to come in for an orientation session at which consent will be obtained. Pregnant smokers will be excluded. They will visit the clinic weekly for 2 months and once monthly for 4 months for a total of 6 months participation.

At each visit they will drink 5 ml of 50:50 ethanol:water containing 10 ug [D10]phenanthrene. They will then collect their 24h urine and return it to the clinic. The urine will be analyzed for [D10]phenanthrene tetraol. The goal of the study is to determine the longitudinal stability of the amount of [D10]phenanthrene-tetraol in urine.

ELIGIBILITY:
Inclusion Criteria:

* smokers and non-smokers
* smoking at least 10 cigarettes daily for the past year (for smokers)
* in good physical health (no unstable medical condition)
* stable, good mental health (not currently, within past 6 months, experiencing unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria).

Exclusion Criteria:

* subjects who have, within the past 6 months, experienced unstable or untreated psychiatric diagnoses, including substance abuse, as determined by the DSM-IV criteria.
* subjects using any other tobacco or nicotine products.
* female subjects who are pregnant or nursing.
* subjects with an unstable medical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 36 hours post dosing
  Deuterated phenanthrene tetraol ([D10]PheT) assessed post dosing for smoked versus oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Hecht, Ph.D., Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (1):
- Tobacco Use Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] ATSDR (Agency for Toxic Substances and Disease Registry). 1990. Toxicological Profile for Polycyclic Aromatic Hydrocarbons. Acenaphthene, Acenaphthylene, Anthracene, Benzo(a)anthracene, Benzo(a)pyrene, Benzo(b)fluoranthene, Benzo(g,i,h)perylene, Benzo(k)fluoranthene, Chrysene, Dibenzo(a,h)anthracene, Fluoranthene, Fluorene, Indeno(1,2,3-c,d)pyrene, Phenanthrene, Pyrene. Prepared by Clement International Corporation, under Contract No. 205-88-0608. ATSDR/TP-90-20.
- [Background] Bock, F.G. and T.L. Dao. 1961. Factors affecting the polynuclear hydrocarbon level in rat mammary glands. Cancer Res. 21: 1024-1029.
- [Background] BOYLAND E, SIMS P. Metabolism of polycyclic compounds. 21. The metabolism of phenanthrene in rabbits and rats: dihydrodihydroxy compounds and related glucosiduronic acids. Biochem J. 1962 Sep;84(3):571-82. doi: 10.1042/bj0840571. No abstract available. PMID 13872198
- [Background] BOYLAND E, WOLF G. Metabolism of polycyclic compounds. 6. Conversion of phenanthrene into dihydroxydihydrophenanthrenes. Biochem J. 1950 Jun-Jul;47(1):64-9. doi: 10.1042/bj0470064. No abstract available. PMID 14791307
- [Background] Budavari, S., M.J. O'Neil and A. Smith (Eds.). 1989. The Merck Index. Merck & Co., Inc. Rahway, NJ, pp. 1143-1144.
- [Background] Buening MK, Levin W, Karle JM, Yagi H, Jerina DM, Conney AH. Tumorigenicity of bay-region epoxides and other derivatives of chrysene and phenanthrene in newborn mice. Cancer Res. 1979 Dec;39(12):5063-8. No abstract available. PMID 498133
- [Background] Chang, L.H. 1943. The fecal excretion of polycyclic hydrocarbons following their administration to the rat. J.. biol. Chem. 151: 93-99.
- [Background] Chaturapit S, Holder GM. Studies on the hepatic microsomal metabolism of (14C) phenanthrene. Biochem Pharmacol. 1978;27(14):1865-71. doi: 10.1016/0006-2952(78)90034-5. No abstract available. PMID 708468
- [Background] FALK HL, KOTIN P, THOMPSON S. INHIBITION OF CARCINOGENESIS. THE EFFECT OF HYDROCARBONS AND RELATED COMPOUNDS. Arch Environ Health. 1964 Aug;9:169-79. doi: 10.1080/00039896.1964.10663816. No abstract available. PMID 14155051
- [Background] GRANT G, ROE FJ. THE EFFECT OF PHENANTHRENE ON TUMOUR INDUCTION BY 3,4-BENZOPYRENE ADMINISTERED TO NEWLY BORN MICE. Br J Cancer. 1963 Jun;17(2):261-5. doi: 10.1038/bjc.1963.37. No abstract available. PMID 14042727
- [Background] HUGGINS C, YANG NC. Induction and extinction of mammary cancer. A striking effect of hydrocarbons permits analysis of mechanisms of causes and cure of breast cancer. Science. 1962 Jul 27;137(3526):257-62. doi: 10.1126/science.137.3526.257. No abstract available. PMID 14449781
- [Background] Polynuclear aromatic compounds, Part 1, Chemical, environmental and experimental data. IARC Monogr Eval Carcinog Risk Chem Hum. 1983 Dec;32:1-453. No abstract available. PMID 6586639
- [Background] Kennaway, E.L. 1924. On the cancer-producing tars and tar-fractions. J. Ind. Hyg. 5: 462-488.
- [Background] LaVoie EJ, Tulley-Freiler L, Bedenko V, Hoffman D. Mutagenicity, tumor-initiating activity, and metabolism of methylphenanthrenes. Cancer Res. 1981 Sep;41(9 Pt 1):3441-7. PMID 7020927
- [Background] Mabey, W.R., J.H. Smith, R.T. Podoll, et al. 1982. Aquatic fate process data for organic priority pollutants. U.S. Environmental Protection Agency, Office of Water Regulations and Standards, Washington, D.C. EPA 440/4-81-014.
- [Background] Nordqvist M, Thakker DR, Vyas KP, Yagi H, Levin W, Ryan DE, Thomas PE, Conney AH, Jerina DM. Metabolism of chrysene and phenanthrene to bay-region diol epoxides by rat liver enzymes. Mol Pharmacol. 1981 Jan;19(1):168-78. No abstract available. PMID 7207460
- [Background] Nousiainen U, Torronen R, Hanninen O. Differential induction of various carboxylesterases by certain polycyclic aromatic hydrocarbons in the rat. Toxicology. 1984 Sep 14;32(3):243-51. doi: 10.1016/0300-483x(84)90077-5. PMID 6089379
- [Background] Pfeiffer EH. Oncogenic interaction of carcinogenic and non-carcinogenic polycyclic aromatic hydrocarbons in mice. IARC Sci Publ (1971). 1977;(16):69-77. PMID 68911
- [Background] Rahman A, Barrowman JA, Rahimtula A. The influence of bile on the bioavailability of polynuclear aromatic hydrocarbons from the rat intestine. Can J Physiol Pharmacol. 1986 Sep;64(9):1214-8. doi: 10.1139/y86-205. PMID 3096546
- [Background] ROE FJ. Effect of phenanthrene on tumour-initiation by 3,4-benzopyrene. Br J Cancer. 1962 Sep;16(3):503-6. doi: 10.1038/bjc.1962.58. No abstract available. PMID 13982333
- [Background] Roe, F.J.C. and G.A. Grant. 1964. Tests of pyrene and phenanthrene for incomplete carcinogenic and anticarcinogenic activity. Br. Emp. Cancer Campaign 41: 59-60. (Abstract) (Cited in IARC, 1983)
- [Background] RTECS (Registry of Toxic Effects of Chemical Substances). 1993. Computer printout.
- [Background] ROE FJ, SALAMAN MH. Further tests for tumour-initiating activity: N, N-di-(2-chloroethyl)-p-aminophenylbutyric acid (CB1348) as an initiator of skin tumour formation in the mouse. Br J Cancer. 1956 Jun;10(2):363-78. doi: 10.1038/bjc.1956.42. No abstract available. PMID 13364128
- [Background] Salamone, M.F. 1981. Toxicity of 41 carcinogenic analogs. Prog. Mutat. Res. 1: 682-685. (Cited in U.S. EPA, 1988)
- [Background] Sax, N.I. and R.L. Lewis (Eds.). 1987. Hawley's Condensed Chemical Dictionary, 11th ed. Van Nostrand Reinhold Company, New York, p. 895.
- [Background] Scribner JD. Tumor initiation by apparently noncarcinogenic polycyclic aromatic hydrocarbons. J Natl Cancer Inst. 1973 Jun;50(6):1717-9. doi: 10.1093/jnci/50.6.1717. No abstract available. PMID 4123924
- [Background] Simmon VF, Rosenkranz HS, Zeiger E, Poirier LA. Mutagenic activity of chemical carcinogens and related compounds in the intraperitoneal host-mediated assay. J Natl Cancer Inst. 1979 Apr;62(4):911-8. PMID 372659
- [Background] Sims P. Qualitative and quantitative studies on the metabolism of a series of aromatic hydrocarbons by rat-liver preparations. Biochem Pharmacol. 1970 Mar;19(3):795-818. doi: 10.1016/0006-2952(70)90243-1. No abstract available. PMID 5507686
- [Background] STEINER PE. Carcinogenicity of multiple chemicals simultaneously administered. Cancer Res. 1955 Oct;15(9):632-5. No abstract available. PMID 13261089
- [Background] Storer JS, DeLeon I, Millikan LE, Laseter JL, Griffing C. Human absorption of crude coal tar products. Arch Dermatol. 1984 Jul;120(7):874-7. PMID 6732260
- [Background] U.S. EPA (U.S. Environmental Protection Agency). 1987. Health and Environmental Effects Profile for Phenanthrene. Prepared by the Environmental Criteria and Assessment Office, Office of Health